CLINICAL TRIAL: NCT04920045
Title: A Trial Comparing a Liberal Versus Restrictive Red Blood Cell Transfusion Strategy on Fatigability, Fatigue, and Activity Levels After Discharge in Hospitalized Patients With Anemia.
Brief Title: A Trial to Assess the Effect of Transfusion Strategies on Fatigability Levels After Hospital Discharge
Acronym: EToF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical practice has shifted such that physician equipoise is lacking, stultifying this study's enrollment. While the scientific question remains relevant, data collection and analysis are complete, and no further research activities are planned.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-0854
Record Dates: First submitted 2021-05-24; First posted 2021-06-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Anemia; Red Blood Cell Transfusion; Fatigability; Fatigue; Physical Function
MeSH Terms: conditions — Anemia; Fatigue | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Intervention Model Description: Randomization will occur after patients have consented to participate and will be done using permuted block de-sign with random blocks of 2, 4, or 6 patients per block.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal Transfusion Arm (Active Comparator): Patient's in the liberal transfusion arm will receive a 1 unit RBC transfusion following randomization and will re-ceive blood in additional 1 unit increments until their Hb is above 9g/dL. At any point during the patient's hospital-ization if their Hb subsequently falls below 9g/dL, they will again be transfused to maintain a Hb>9g/dL, and this will be maintained throughout their hospitalization.
  Interventions: Other: Red blood cell transfusion
- Restrictive Transfusion Arm (Active Comparator): Patients in the restrictive transfusion arm will receive transfusion if their Hb concentration falls below 7g/dL. RBC's will be administered 1 unit at a time and enough blood will be given to increase patient's Hb to above 7g/dL.
  Interventions: Other: Red blood cell transfusion

INTERVENTIONS:
Other: Red blood cell transfusion — All RBC transfusions will be administered in 1 unit increments to maintain patients' Hb concentration above the trial arm threshold they are randomized to. All transfusions will be followed by a Hb measure and an additional unit(s) of RBC's will only be transfused if there is documentation of the patient's Hb concentration below the trial arm threshold they are randomized to. However, in the case of life-threatening bleeding clinicians will be able to transfuse patients without first checking a patient's Hb concentration. Once randomized, patients will be man-aged according to protocol until hospital discharge independent of transfer to another service and/or specialized hospital ward.

SUMMARY:
This study is a randomized controlled trial in which hospitalized patients with anemia are randomized to receive transfusion at: a) Hb<9g/dL (liberal transfusion strategy), or b) Hb<7g/dL (restrictive transfusion strategy). We are measuring self-reported fatigability, fatigue, and activity levels at randomization and 7 days post hospital discharge in both trial arms. In a subset of 75 patients in each trial arm (150 total), we will are administering the 6 Minute Walk Test at randomization and 7 days post discharge.

DETAILED DESCRIPTION:
The design of this proposed study is a randomized controlled trial of hospitalized adult general medicine patients with anemia at the University of Chicago (UC). Patients will be randomized to receive transfusion at either a hemoglobin (Hb)<9g/dL (liberal arm) or a Hb<7g/dL (restrictive arm) throughout their hospitalization. Self-reported fatigability, fatigue, and activity levels will be measured in consented patients at randomization and through a follow-up phone call 7 days after hospital discharge. We will also enroll 150 patients to participate in the Six Minute Walk Test85,86 (6MWT) at randomization and in the clinic 7 days after hospital discharge.

This trial will test whether a liberal transfusion strategy is superior to a restrictive transfusion in hospitalized patients with anemia on fatigability levels after hospital discharge. Our primary outcome is self-reported fatigability level 7 days after hospital discharge measured using the Pittsburgh Fatigability Scale (PFS)71. Secondary outcomes include fatigue measured using the Patient Reported Outcome Measurement Information System (PROMIS) Fatigue Aa instrument, and activity measured by the Physical Activity Scale for the Elderly, and 6MWT distance.

Eligible patients for this trial will be recruited from the University of Chicago Medical Center (UCMC) general medicine services using the University of Chicago Hospitalist Project (UCHP) research infrastructure. The eligibility criteria is: 1) hospitalized adult >18 years of age, 2) admitted to the general medicine services at the University of Chicago, 3) any Hb concentration of <9g/dL during their hospitalization. We will exclude patients who: 1) decline blood transfusion, 2) and/or who have a diagnosis of sickle cell anemia, 3) and/or are brain dead or receiving only palliative treatment, 4) and/or are unable to follow-up after discharge. We will not exclude patients who received transfusion prior to randomization. Eligible patients will be identified using the encrypted UCHP research database, which is programmed to extract real time EHR data into the database in order to identify patients potentially eligible for participation in research studies. The PI and Study Coordinator (SC) will be responsible for patient recruitment and consent.

Consenting patients will be randomized to either receive transfusion when their Hb drops below 7g/dL (restrictive arm) or 9g/dl (liberal arm) at any point during hospitalization, and randomized assignment will be done using permuted block design with random blocks of 2, 4, or 6 patients per block. All red blood cell (RBC) transfusions will be administered in 1 unit increments in order to maintain patients' Hb concentration above the trial arm threshold they are randomized to. All transfusions will be followed by a Hb measure and an additional unit(s) of RBC's will only be transfused if there is documentation of the patient's Hb concentration below the trial arm threshold they are randomized to. However, In the case of life-threatening bleeding clinicians will be free to transfuse patients without first checking a patient's Hb concentration. Once randomized, patient's will be managed according to protocol until hospital discharge independent of transfusion to another service and/or specialized hospital ward. This trial will not control or dictate transfusion of other blood products, which will be administered at the discretion of the attending physician caring for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized on a general medicine service at the University of Chicago
* Any hemoglobin (Hb) concentration <9g/dL

Exclusion Criteria:

* Have sickle cell anemia
* Decline blood transfusion
* Are receiving palliative care treatment only
* Are brain dead
* Cannot follow up after hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Change in self-reported fatigability level | Fatigability will be measured at admission to the hospital during the index hospitalization and 7 days after hospital discharge.
  Self-reported fatigability will be measured by the Pittsburgh Fatigability Scale (PFS). The PFS is a 10 item scale that ranges from 0-50 with greater scores indicating greater fatigability.

SECONDARY OUTCOMES:
Change in self-reported fatigue level | Fatigue will be measured at admission to the hospital during the index hospitalization and 7 days after hospital discharge.
  Self-reported fatigue will be measured by the Patient-Reported Outcome Measurement Information System (PROMIS-F) Fatigue 8a instrument.The PROMIS-F scores range from 8-40, with higher scores indicating greater fatigue.
Change in self-reported activity level | Activity will be measured at admission to the hospital during the index hospitalization and 7 days after hospital discharge.
  Self-reported activity will be measure by the Physical Activity Scale for the Elderly (PASE). Higher scores on the PASE indicated greater physical activity.
Change in 6 Minute Walk Test (6MWT) distance | 6MWT will be measured at admission to the hospital during the index hospitalization and 7 days after hospital discharge.
  6MWT is measure of functional capacity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066